CLINICAL TRIAL: NCT03965039
Title: A Randomized Clinical Study to Assess the Effects of Various Dentifrice Technologies on Dentinal Hypersensitivity
Brief Title: A Clinical Study to Assess the Effects of Various Dentifrice Technologies on Dentinal Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019079
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Results first posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Marketed stannous fluoride toothpaste (Active Comparator): Brush twice daily
  Interventions: Drug: Stannous fluoride toothpaste
- Marketed potassium nitrate toothpaste (Active Comparator): Brush Twice Daily
  Interventions: Drug: Potassium nitrate toothpaste
- Marketed sodium monofluorophosphate toothpaste (Placebo Comparator): Brush Twice Daily
  Interventions: Drug: Sodium monofluorophosphate toothpaste
- Experimental dipotassium oxalate toothpaste (Experimental): Brush Twice Daily
  Interventions: Device: Dipotassium oxalate toothpaste

INTERVENTIONS:
Device: Dipotassium oxalate toothpaste — Experimental dipotassium oxalate (3%) toothpaste
  Arms: Experimental dipotassium oxalate toothpaste
Drug: Stannous fluoride toothpaste — Marketed stannous fluoride (0.454%) toothpaste
  Arms: Marketed stannous fluoride toothpaste
Drug: Potassium nitrate toothpaste — Marketed potassium nitrate (5%) toothpaste
  Arms: Marketed potassium nitrate toothpaste
Drug: Sodium monofluorophosphate toothpaste — Marketed sodium monofluorophosphate (0.76%) toothpaste
  Arms: Marketed sodium monofluorophosphate toothpaste

SUMMARY:
The objective of this study is to evaluate the efficacy (changes in dentinal hypersensitivity) and safety (oral soft tissue evaluation) after use of one of four dentifrices in subjects with pre-existing hypersensitivity over an 11-week period.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age;
* provide written informed consent prior to participation and be given a signed copy of the informed consent form;
* sign a Confidentiality Disclosure Agreement (CDA);
* be in good general health as determined by the Investigator/designee;
* agree not to participate in any other oral/dental product studies during the course of this study;
* agree to delay any dentistry (including dental prophylaxis) until the study has been completed;
* agree to refrain from the use of any non-study oral hygiene products*;
* exhibit adequate oral hygiene (i.e., brush teeth daily and exhibit no signs of oral neglect);
* have an absence of extensive calculus above the gum line;
* agree to return for all scheduled visits and follow study procedures; and
* have two teeth with a Schiff sensitivity score > 1 in response to air challenge and a Yeaple probe score of 10-20 g in response to tactile challenge. (If these two eligible teeth are located in the same quadrant, they have to be separated by 2 other teeth.)

Exclusion Criteria:

* having taken anti-inflammatory, analgesic, or psychotropic drugs, chronically;
* chronic medical debilitating disease associated with constant or intermittent episodes of daily pain;
* any home-care bleaching, whitening products or have had a professional bleaching treatment within 4 weeks of the Baseline visit;
* dental prophylaxis within 2 weeks prior to Baseline visit;
* having received professional desensitizing treatment or having used over-the-counter desensitizing products within 6 weeks of the Baseline visit;
* having periodontal surgery, orthodontic treatment, or teeth restored in the preceding three months;
* having teeth or periodontium with pathology or defects likely to cause pain;
* having a history of allergies or hypersensitivity to ingredients in commercial dental products or cosmetics;
* self-reported pregnancy or lactation;
* having self-reported eating disorders, uncontrolled gastroesophageal reflux disease (GERD or Acid Reflux), excessive dietary or environmental exposure to acids, or other systemic conditions that are predisposing to dentinal hypersensitivity;
* history or presence of kidney disorders, kidney stones, have celiac disease, inflammatory bowel disease (ulcerative colitis or Crohn's disease), chronic pancreatitis, have had intestinal or weight-loss surgery, or if have stomach or intestinal problems that keep them from absorbing certain foods or nutrients;
* any diseases or condition that might interfere with the safe participation in the study;
* inability to undergo study procedures;
* having severe xerostomia;
* having had active caries within the 12 months;
* having high risk for caries development (rampant caries, multiple dental restorations, crowns with compromised margin) per examiners discretion;
* teeth will be excluded from study measurements if they:

  * have deep, defective, or facial restorations;
  * have full crowns, extensive caries, cracked enamel, or are abutment teeth for fixed or removable prosthesis;
  * present with tendency for spontaneous bleeding;
  * have been scaled/root planed or restored within the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Silverstone Research Group, Las Vegas, Nevada, United States

REFERENCES:
- [Derived] Biesbrock AR, He T, Zou Y, Grender JM, Amini P, Sagel PA, Groth A, Klukowska M. Randomized clinical trial evaluating kinetic benefits of desensitizing agents: Magnitude, onset, and stability of relief. J Periodontol. 2025 May 30. doi: 10.1002/JPER.24-0688. Online ahead of print. PMID 40444818

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Marketed Stannous Fluoride Toothpaste | Marketed Potassium Nitrate Toothpaste | Marketed Sodium Monofluorophosphate Toothpaste | Experimental Dipotassium Oxalate Toothpaste
Started | 30 | 30 | 30 | 30
Completed | 30 | 29 | 30 | 29
Not Completed | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Marketed Stannous Fluoride Toothpaste | Marketed Potassium Nitrate Toothpaste | Marketed Sodium Monofluorophosphate Toothpaste | Experimental Dipotassium Oxalate Toothpaste | Total
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.73 (11.52) | 42.53 (13.28) | 39.03 (11.04) | 39.87 (10.42) | 40.04 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 21 | 22 | 86
  Male | 8 | 9 | 9 | 8 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 6 | 7 | 25
  Not Hispanic or Latino | 25 | 23 | 24 | 23 | 95
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 5 | 1 | 2 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 3 | 2 | 7 | 7 | 19
  White | 20 | 24 | 15 | 15 | 74
  More than one race | 1 | 3 | 5 | 7 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Air Challenge
Description: The Schiff Sensitivity Scale will be assessed for each test tooth via an evaporative air challenge. The examiner will record the Schiff Index score corresponding to the response to the air challenge. The Schiff Index Sensitivity scale is scored as follows- 0: tooth/subject did not respond to stimulus, 1: tooth/subject responds to stimulus, but does not request discontinuation of stimulus, 2: tooth/subject responds to stimulus and requests discontinuation or moves form stimulus, 3: tooth/subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. The higher the Schiff score, the more sensitive the tooth. The least square mean will be calculated for this measure.
Time Frame: 4 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Marketed Stannous Fluoride Toothpaste | Marketed Potassium Nitrate Toothpaste | Marketed Sodium Monofluorophosphate Toothpaste | Experimental Dipotassium Oxalate Toothpaste
Number analyzed (Participants) | 30 | 30 | 30 | 28
score on a scale | 1.17 (0.141) | 1.48 (0.087) | 2.26 (0.066) | 1.39 (0.116)

2. Secondary Outcome: Baseline Air Challenge
Description: The Schiff Sensitivity Scale will be assessed for each test tooth via an evaporative air challenge. The examiner will record the Schiff Index score corresponding to the response to the air challenge. The Schiff Index Sensitivity scale is scored as follows- 0: tooth/subject did not respond to stimulus, 1: tooth/subject responds to stimulus, but does not request discontinuation of stimulus, 2: tooth/subject responds to stimulus and requests discontinuation or moves form stimulus, 3: tooth/subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. The higher the Schiff score, the more sensitive the tooth.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Marketed Stannous Fluoride Toothpaste | Marketed Potassium Nitrate Toothpaste | Marketed Sodium Monofluorophosphate Toothpaste | Experimental Dipotassium Oxalate Toothpaste
Number analyzed (Participants) | 30 | 30 | 30 | 30
score on a scale | 2.45 (0.379) | 2.40 (0.381) | 2.52 (0.382) | 2.45 (0.356)

3. Secondary Outcome: Air Challenge
Description: as for outcome 1
Time Frame: 3 days
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Marketed Stannous Fluoride Toothpaste | Marketed Potassium Nitrate Toothpaste | Marketed Sodium Monofluorophosphate Toothpaste | Experimental Dipotassium Oxalate Toothpaste
Number analyzed (Participants) | 30 | 30 | 29 | 30
score on a scale | 1.93 (0.081) | 2.05 (0.085) | 2.36 (0.062) | 1.88 (0.085)

4. Secondary Outcome: Air Challenge
Description: as for outcome 1
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Marketed Stannous Fluoride Toothpaste | Marketed Potassium Nitrate Toothpaste | Marketed Sodium Monofluorophosphate Toothpaste | Experimental Dipotassium Oxalate Toothpaste
Number analyzed (Participants) | 30 | 30 | 30 | 29
score on a scale | 1.44 (0.117) | 1.78 (0.092) | 2.24 (0.074) | 1.61 (0.103)

5. Secondary Outcome: Air Challenge
Description: as for outcome 1
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Marketed Stannous Fluoride Toothpaste | Marketed Potassium Nitrate Toothpaste | Marketed Sodium Monofluorophosphate Toothpaste | Experimental Dipotassium Oxalate Toothpaste
Number analyzed (Participants) | 30 | 29 | 30 | 29
score on a scale | 0.96 (0.144) | 1.24 (0.094) | 2.22 (0.059) | 1.18 (0.134)

6. Secondary Outcome: Air Challenge
Description: The Schiff Sensitivity Scale will be assessed for each test tooth via an evaporative air challenge. The examiner will record the Schiff Index score corresponding to the response to the air challenge. The Schiff Index Sensitivity scale is scored as follows- 0: tooth/subject did not respond to stimulus, 1: tooth/subject responds to stimulus, but does not request discontinuation of stimulus, 2: tooth/subject responds to stimulus and requests discontinuation or moves form stimulus, 3: tooth/subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. The higher the Schiff score, the more sensitive the tooth. The least square mean will be calculated for this measure. All subjects will have been on three weeks use of a marketed sodium monofluophosphate toothpaste (from week 8 to week 11).
Time Frame: 11 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Marketed Stannous Fluoride Toothpaste | Marketed Potassium Nitrate Toothpaste | Marketed Sodium Monofluorophosphate Toothpaste | Experimental Dipotassium Oxalate Toothpaste
Number analyzed (Participants) | 30 | 29 | 30 | 29
score on a scale | 1.32 (0.147) | 1.40 (0.121) | 2.18 (0.071) | 1.32 (0.145)

7. Secondary Outcome: Baseline Yeaple Probe
Description: Tactile Threshold will be measured using a Yeaple probe. Testing is performed beginning at 10 g. The examiner records tactile scores for responding teeth. After treatment, testing begins at 10 g and increases by 10 g to a maximum of 50 g. The higher the tactile threshold, the less sensitive the tooth. Each successive challenge increases until a "yes" response is repeated. If a second "yes" is not obtained, the force setting is increased to the next step and continued until a force is found which elicits two consecutive "yes" responses and will be recorded as the threshold on the Tactile Sensitivity Score form.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Marketed Stannous Fluoride Toothpaste | Marketed Potassium Nitrate Toothpaste | Marketed Sodium Monofluorophosphate Toothpaste | Experimental Dipotassium Oxalate Toothpaste
Number analyzed (Participants) | 30 | 30 | 30 | 30
score on a scale | 10.33 (1.826) | 10.50 (1.526) | 11.00 (2.754) | 10.50 (2.013)

8. Secondary Outcome: Tactile Threshold
Description: Tactile Threshold will be measured using a Yeaple probe. Testing is performed beginning at 10 g. The examiner records tactile scores for responding teeth. After treatment, testing begins at 10 g and increases by 10 g to a maximum of 50 g. The higher the tactile threshold, the less sensitive the tooth. Each successive challenge increases until a "yes" response is repeated. If a second "yes" is not obtained, the force setting is increased to the next step and continued until a force is found which elicits two consecutive "yes" responses and will be recorded as the threshold on the Tactile Sensitivity Score form. The least square mean will be calculated for this measure.
Time Frame: 3 days
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Marketed Stannous Fluoride Toothpaste | Marketed Potassium Nitrate Toothpaste | Marketed Sodium Monofluorophosphate Toothpaste | Experimental Dipotassium Oxalate Toothpaste
Number analyzed (Participants) | 30 | 30 | 29 | 30
score on a scale | 16.70 (1.039) | 13.74 (0.704) | 12.41 (0.741) | 15.90 (1.240)

9. Secondary Outcome: Tactile Threshold
Description: as for outcome 8
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Marketed Stannous Fluoride Toothpaste | Marketed Potassium Nitrate Toothpaste | Marketed Sodium Monofluorophosphate Toothpaste | Experimental Dipotassium Oxalate Toothpaste
Number analyzed (Participants) | 30 | 30 | 30 | 29
score on a scale | 22.70 (1.987) | 18.57 (1.528) | 14.17 (1.022) | 21.61 (1.533)

10. Secondary Outcome: Tactile Threshold
Description: as for outcome 8
Time Frame: 4 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Marketed Stannous Fluoride Toothpaste | Marketed Potassium Nitrate Toothpaste | Marketed Sodium Monofluorophosphate Toothpaste | Experimental Dipotassium Oxalate Toothpaste
Number analyzed (Participants) | 30 | 30 | 30 | 28
score on a scale | 26.76 (2.548) | 22.76 (1.710) | 13.93 (0.988) | 25.06 (1.556)

11. Secondary Outcome: Tactile Threshold
Description: as for outcome 8
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Marketed Stannous Fluoride Toothpaste | Marketed Potassium Nitrate Toothpaste | Marketed Sodium Monofluorophosphate Toothpaste | Experimental Dipotassium Oxalate Toothpaste
Number analyzed (Participants) | 30 | 29 | 30 | 29
score on a scale | 29.30 (2.728) | 27.45 (1.926) | 13.45 (0.824) | 28.49 (2.044)

12. Secondary Outcome: Tactile Threshold
Description: Tactile Threshold will be measured using a Yeaple probe. Testing is performed beginning at 10 g. The examiner records tactile scores for responding teeth. After treatment, testing begins at 10 g and increases by 10 g to a maximum of 50 g. The higher the tactile threshold, the less sensitive the tooth. Each successive challenge increases until a "yes" response is repeated. If a second "yes" is not obtained, the force setting is increased to the next step and continued until a force is found which elicits two consecutive "yes" responses and will be recorded as the threshold on the Tactile Sensitivity Score form. The least square mean will be calculated for this measure. All subjects will have been on three weeks use of a marketed sodium monofluorophosphate toothpaste (from week 8 to week 11).
Time Frame: 11 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Marketed Stannous Fluoride Toothpaste | Marketed Potassium Nitrate Toothpaste | Marketed Sodium Monofluorophosphate Toothpaste | Experimental Dipotassium Oxalate Toothpaste
Number analyzed (Participants) | 30 | 29 | 30 | 29
score on a scale | 24.75 (2.631) | 21.92 (1.801) | 12.71 (0.664) | 24.85 (1.863)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for all 11 weeks of the study for each intervention.
Arm/Group | Marketed Stannous Fluoride Toothpaste | Marketed Potassium Nitrate Toothpaste | Marketed Sodium Monofluorophosphate Toothpaste | Experimental Dipotassium Oxalate Toothpaste
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 5/30 | 0/30 | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Marketed Stannous Fluoride Toothpaste (N=30) | Marketed Potassium Nitrate Toothpaste (N=30) | Marketed Sodium Monofluorophosphate Toothpaste (N=30) | Experimental Dipotassium Oxalate Toothpaste (N=30)
Desquamation Mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Mouth Injury (Gastrointestinal disorders) | 0 | 4 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI should disclose plans to sponsor prior to public release.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/39/NCT03965039/Prot_SAP_000.pdf